CLINICAL TRIAL: NCT04092205
Title: EMERA007 - An Open Label, Active-treatment Controlled, Phase 2a Pilot Study to Explore Safety and Efficacy of NBMI Treatment in Patients With Beta Thalassemia Major, Requiring Iron Chelation
Brief Title: Phase 2a Pilot Study of NBMI Treatment in Patients With Beta Thalassemia Major, Requiring Iron Chelation
Acronym: EMERA007
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EmeraMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMERA007
Record Dates: First submitted 2019-07-29; First posted 2019-09-17 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — N,N'-Bis(2-mercaptoethyl)isophthalamide

STUDY DESIGN:
Intervention Model Description: An open label, active-treatment controlled once daily oral administration for 28 days and 28 days follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Treatment (Experimental): 28 days treatment with NBMI 600 mg/day
  Interventions: Drug: Emeramide

INTERVENTIONS:
Drug: Emeramide — Lipophilic, membrane passing Metal chelator and anti oxidant
  Other Names: NBMI; Irminix

SUMMARY:
A pilot study to explore safety and efficacy of NBMI treatment in patients with Beta Thalassemia Major requiring iron chelation

Investigational product: NBMI (N1,N3-bis(2-mercaptoethyl) isophthalamide), INN: Emeramide

Indication: Beta Thalassemia Major

DETAILED DESCRIPTION:
Patients with iron overload, not controlled with current therapy will be enrolled to the study. After initial treatment with standard chelation therapy (deferasirox), patients will receive 600 mg daily dose of emeramide (NBMI) for 28 days. After that follow up period on standard treatment with deferasirox shall follow.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has clinically confirmed documented diagnosis of Beta Thalassemia Major, according to the current clinical criteria, and are on blood transfusions.
2. Patient has been on a stable maintaince therapy with deferasirox for at least during last 3 months.
3. Patients current chelation therapy is considered inadequate, meaning that there is evidence from clinical monitoring that chronic iron overload is present (e.g. serum ferritin >1,000 µg/l), for at least during the last 3 months.
4. The ferritin level has been stable with max 10% difference between max-to-low, and the iron chelator treatment dose has been unchanged during the last 3 months
5. Patient is aged 18 years or older at screening.
6. Female patients are only eligible for the study if they are either surgically sterile or at least 2 years postmenopausal, or have a negative result of serum hCG test at screening and if willing to use acceptable, effective methods of contraception during the trial and for three month after the end of trial participation as defined inpoint 7.7. of this the protocol.
7. Male patients must either be surgically sterile or he and his female spouse/partner who is of childbearing potential must be willing to use highly effective methods of contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continuing throughout the study.
8. Patient is fluent in the local language and provides written informed consent.

Exclusion Criteria:

1. Known history or presence of clinically significant other, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Known or suspected allergy hypersensitivity or idiosyncratic reaction to NBMI or any other drug substances with similar activity.
3. History of drug or alcohol addiction requiring treatment.
4. History of malabsorption within the last year or presence of clinically significant gastrointestinal disease or surgery that may affect drug bioavailability, including but not limited to cholecystectomy.
5. Presence of hepatic or renal dysfunction. (SGOT and SGPT and bilirubin > X3 (3 fold) UNL. creatinine > 1.5mg/dl).
6. Female patient who is pregnant (serum hCG level consistent with pregnancy diagnosis); or breastfeeding.
7. Participation in a clinical trial that involved administration of an investigational medicinal product within 90 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
8. Have clinically significant abnormal laboratory values (e.g. liver enzymes).
9. Have clinically significant findings from a physical examination (e.g. fever).
10. Patient has Inflammatory disorders, liver disease such as hepatitis, malignancy or other condition that could influence ferritine levels and therefore validity of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  The safety assessment is based on the number, type and severity of adverse events. The incidence of adverse events will be summarized by organ class, severity and duration.

SECONDARY OUTCOMES:
Change in serum ferritin levels | 28 days
  Change in serum ferritin levels measured in µg/l (V2 level compared to V4 level and V5 level compared to V2 level)
Change in iron load in the liver and heart | 28 days
  Change in iron load in the liver and heart as measured by magnetic resonance imaging (MRI) techniques for assessing tissue iron T* (V2 level compared to V4 level and V5 level compared to V2 level)
Percentage of NBMI-treated patients who will develop a response | 28 days
  Percentage of NBMI-treated patients who will develop a response to NBMI (response will be defined as lack of increase of ferritin levels ) as compared between V2 level and V4 level

OTHER OUTCOMES:
Kidney markers (serum creatinine levels, glomerular filtration calculation) | 28 days
  Change from baseline after both treatments. Serum creatinine levels will be measured in μmol/l, glomerular filtration in ml/min.
Pharmacokinetic parameters | Visit 4, 5, 6, 7
  Pharmacokinetic parameters derived from plasma concentrations of NBMI (Time of maximum analyte concentration - Tmax, Maximum drug concentration - Cmax,The terminal elimination rate constant - λz, Apparent terminal elimination half-life - t1/2, The area under the plasma concentration - AUC0-t, Area under the concentration-time curve - AUC0-∞, Area under the concentration-time curve - AUC%Extrap)
Malondialdehyde levels | Visit 2, 4
  Indicator of oxidative stress measured in μmol/l.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center "Mother Theresa" Tirana, Tirana, Albania

IPD SHARING:
Plan to Share IPD: No